CLINICAL TRIAL: NCT04645992
Title: Effect Yoga in Addition to TENS on Diabetic Glaucoma
Brief Title: Effect of Combining Yoga to TENS on Diabetic Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002604
Record Dates: First submitted 2020-11-21; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus; Glaucoma
MeSH Terms: conditions — Diabetes Mellitus; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): study group will receive only one session of yoga eye exercise for 20 minutes followed by transcutaneous electrical nerve stimulation by placing electrodes on skin over urinary bladder (BL) acupoints 61 and 62 for 20 minutes
  Interventions: Device: active TENS
- control group (Sham Comparator): control group will be treated with the same protocol as the study group but with the unit of transcutaneous electrical nerve stimulation is off .
  Interventions: Device: sham TENS

INTERVENTIONS:
Device: active TENS — study group will receive only one session of yoga eye exercise for 20 minutes followed by TENS by placing electrodes on skin over urinary bladder (BL) acupoints 61 and 62 for 20 minutes
  Arms: study group
Device: sham TENS — control group will be treated with the same protocol as the study group but with the TENS unit is off .
  Arms: control group

SUMMARY:
Intraocular pressure (IOP) is maintained by a balance between aqueous production and outflow with an imbalance leading to elevated eye pressure. Very high levels of IOP will subject retinal cells to mechanical stress. In addition to mechanical injury, IOP elevation can impair ocular blood flow reducing perfusion pressure to retinal neurons. Long-term vascular and mechanical stresses can produce further injury at the optic nerve.

Elevated intraocular pressure (IOP) or ocular hypertension (OHT) is the only well-established modifiable risk factor for primary open-angle glaucoma (POAG), the most common form of glaucoma. Glaucoma is a class of optic neuropathy. It is main leading cause of blindness.

Glaucoma is classified on the basis of anatomic features as open angle (where the anterior chamber angle of the eye remains open) and angle-closure (with closure of the anterior chamber angle). Glaucoma is considered primary if the eye has no preexisting disease. Secondary forms of glaucoma are caused by various ocular or systemic diseases such as pigment dispersion syndrome and ocular trauma.

It seems reasonable to consider that a longer duration of diabetes mellitus (DM) with a prolonged insult to the retina and optic nerve via vascular, glial, and neuronal factors would be associated with a higher risk of OAG.

DETAILED DESCRIPTION:
patients with diabetic glaucoma (80 patients ) from both sexes will be divided to 2 groups, 40 patients for each group;

study group will receive only one session of 20 minutes yoga ocular training for 20 minutes followed by transcutaneous electrical nerve stimulation (TENS) by placing electrodes on skin over urinary bladder (BL) acupoints 61 and 62 for 20 minutes

control group will be treated with the same protocol as the study group but with the TENS unit is off.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM duration more than 5 years .
* BMI will be < 30 kg/m² .
* patients with bilateral primary open-angle glaucoma.

Exclusion Criteria:

* acute or chronic eye inflammation
* cataract
* eye surgeries
* mental ill patients
* patients who will refuse to participate in the study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 80 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Intraoccular pressure measurement | immediately after the session
  it will be measured in right and left eye

SECONDARY OUTCOMES:
Intraoccular pressure measurement | immediately after thirty minutes of session
  it will be measured in right and left eye
Intraoccular pressure measurement | immediately after sixty minutes of session end
  it will be measured in right and left eye

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt